CLINICAL TRIAL: NCT01680042
Title: Phase 1 Study of Phenytoin Mucoadhesive Paste for Wound Healing After Oral Biopsy
Brief Title: Clinical Effect of Phenytoin Mucoadhesive Paste on Wound Healing After Oral Biopsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, somayeh alirezaei, resident, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Merck-023
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Wound Healing; Pain
Keywords: inflammatory halo; VAS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phenytoin paste (Active Comparator): this group receives phenytoin paste after oral biopsy
  Interventions: Drug: Phenytoin paste
- usual mucoadhesive paste (Placebo Comparator): this group receives the usual mucoadhesive paste without phenytoin after oral biopsy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenytoin paste
  Arms: phenytoin paste
Drug: Placebo
  Arms: usual mucoadhesive paste

SUMMARY:
several studies have investigated healing effect of phenytoin.In this study we investigate healing effect of phenytoin mucoadhesive paste comparing to the usual mucoadhesive paste after oral biopsy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergone oral biopsy

Exclusion Criteria:

* systemic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
healing biopsy wound | 7 days
  patient recieves phenytoin mucoadhesive paste after oral biopsy and the diameter of inflammatory halo is determined in 1,3,5and the 7th days.pain measurment is also assesed by VAS score

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Shaheed Beheshti University, Tehran
  - Shahid Beheshti Medical University, Tehran